CLINICAL TRIAL: NCT07400978
Title: An At-distance and Online Intervention to Promote Parental Involvement and Self-regulation: Study Protocol for a Cluster Randomized Controlled Trial
Brief Title: An At-distance and Online Intervention to Promote Parental Involvement and Self-regulation
Acronym: Lupis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Sandra Mesquita, Principal Investigator, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEICSH 037/2022; 2021.07428.BD (Other Grant/Funding Number: FCT (Foundation for Science and Technology))
Record Dates: First submitted 2026-01-21; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Parental Involvement; Self-regulation in Children
Keywords: Parental Involvement; Self-regulation; Parental Intervention; At-distance intervention program; Online intervention program
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Intervention Model Description: A three-armed cluster randomized controlled trial will be conducted. It will include: (i) Experimental Group (EG), in this condition for eight weekly modules, parents will be delivered modules about SR strategies (e.g., goal-setting) through a narrative-based intervention program; (ii) Active Control Group (ACG) parents in this condition will benefit during eight weekly modules from general educational content focused on study skills (e.g., making a study timetable); (iii) Passive Control Group (PCG) where parents will not benefit from an intervention.
Who Masked: Participant
Masking Description: We will be conducting a single-blind study, as the nature of the interventions will not allow the implementers to be blinded. The schools and individual participants will, however, be blinded to the group to which they will belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group - At-distance and online intervention across a private Facebook® group. (Experimental): This group will participate in eight modules on self-regulation strategies delivered in an at-distance and online format, which aim to promote parental involvement and, consequently, self-regulation in children. Participants will be parents of students in the first and second years of elementary school.
  Interventions: Behavioral: Lupis program: parental intervention to promote self-regulation in children
- Active Control Group - At-distance and online intervention across a private Facebook® group (Experimental): This group will participate in eight modules on study methods delivered in an at-distance and online format, which aim to promote parental involvement and, consequently, self-regulation in children. Participants will be parents of students in the first and second years of elementary school.
  Interventions: Behavioral: Parental intervention on study methods
- Passive Control Group (No Intervention): This group of parents will not benefit from intervention and will respond to assessment moments.

INTERVENTIONS:
Behavioral: Lupis program: parental intervention to promote self-regulation in children — Narrative-based intervention-the self-regulation strategies covered in each module (e.g., goal setting and asking for help).
  Each module will include: i) a video discussing self-regulation strategies incorporated into "The Three Little Pigs" tale; ii) three activities related to the video content; iii) a weekly synchronous group videoconference session with a trained educational psychologist acting as a mediator.
  Arms: Experimental Group - At-distance and online intervention across a private Facebook® group.
Behavioral: Parental intervention on study methods — Each module will include: i) a video discussing study methods; ii) three activities related to the video content; iii) a weekly synchronous group videoconference session with a trained educational psychologist acting as a mediator.
  Arms: Active Control Group - At-distance and online intervention across a private Facebook® group

SUMMARY:
Parents play a significant role in their children's development and learning. Parental involvement (PI) is characterized by behavioral profiles that are manifested in activities at home (e.g., helping with homework) and school (e.g., participating in meetings with teachers). Involved parents tend to create more opportunities for their children to develop different competencies. These competencies are relevant to children's academic success, namely, the knowledge and use of self-regulation (SR) strategies. SR strategies enable children to take control and responsibility for their behaviors, thoughts, and emotions, thereby achieving a goal (e.g., an academic goal), which in turn leads to higher academic performance and well-being.

Extensive research has identified PI and SR as strong predictors of children's academic success, underscoring the need to promote them actively. Thus, the main goal of this investigation - the Lupis program - is to develop and evaluate the efficacy of an at-distance and online intervention program for parents of 1st and 2nd grade elementary school students. The Lupis will be a narrative-based intervention, utilizing wise intervention techniques in its design. The Lupis program will aim to promote PI and, consequently, SR competencies in children.

In general, it is expected to develop an effective intervention program to promote PI and SR competencies in children. Additionally, Lupis is expected to help parents and children prevent and address the challenges of transitioning from preschool to elementary school with essential competencies for children's learning and academic success.

DETAILED DESCRIPTION:
Parents are primarily responsible for children's development and learning. The communication between parents and children about school, including the expectations and aspirations that parents have for their children, as well as the school's aspects, such as parents' attendance and participation in school activities, is commonly referred to as Parental Involvement (PI). Increased PI in children's lives seems to be positively associated with a positive impact on children's development, particularly in mastery of self-regulation (SR) competencies. SR competencies are a complex process in which individuals take control of and are responsible for their behaviors, cognitions, and emotions in achieving self-established goals. SR behaviors are highly related to inhibitory and attention control when individuals pursue goals. There is thus a relationship with executive functioning, as it is executive functions (EF) that enable the active process of SR to occur.

Parenting literature is unanimous in that the SR is a process influenced by the individual, and therefore, it can be taught and improved through effective parenting. Parental intervention programs emerge as a valuable tool to address and support parents' educational needs. Parents' engagement in these programs increases their competency to help their children's learning process. However, parents' enrollment in in-person programs is challenging (e.g., displacement difficulties, costs, and the availability of courses). To overcome these difficulties, researchers investigated the efficacy of at-distance and online programs. The investigators found that these interventions are effective and allow overcoming barriers, such as lower costs, time flexibility, and easy accessibility.

Typically, interventions for parents are designed to address problem-centered needs (e.g., in language development in children). These programs are usually focused on a particular topic, but they may lose peripheral awareness. It is necessary to develop programs for parents that are not focused on a specific educational problem, but rather preventive programs, addressing everyday problems such as social, emotional, and behavioral issues that parents have to cope with daily.

Thus, this investigation aims to help respond to this need highlighted in the literature, with the main purpose being to develop and evaluate the efficacy of an at-distance and online intervention program (Lupis program) to promote PI and, and influence the development the SR strategies in their children, delivered through Facebook® for parents of children in the 1st and 2nd grades. This purpose arises from the recognition of PI and SR as strong predictors of children's educational trajectory, as it is crucial to promote parents' competencies to help them intervene in the early stages of children's learning.

The Lupis program - Theoretical rationale Lupis is grounded on the Hoover-Dempsey and Sandler model of the PI process, developed by Hoover-Dempsey and Sandler and updated over the years. The model is divided into five main levels, with the two levels referring to what motivates parents to become involved in their children's education (e.g., their perception of self-efficacy - level 1) and how the parents do so (e.g., by using learning mechanisms - level 1.5 and 2). The remaining levels concern how children perceive this PI (level 3) and its impact on their development, particularly in terms of knowledge and use of SR strategies, as well as academic success (levels 4 and 5).

Regarding SR, the framework underlying the Lupis program is social cognitive theory, which explains individual learning as the result of the interaction among personal, behavioral, and environmental factors. The SR model describes how individuals engage in their own learning; it is a cyclical model and consists of three phases (the preliminary phase, the performance or volitional control phase, and the self-reflection phase). Later proposed as the cyclical PLEE model (i.e., Planning, Execution, and Evaluation), where each of these phases of the PLEE process activates a PLEE cycle that takes place within it.

Theoretical tools:

- A narrative-based intervention program using types of knowledge and instructional sequence.

The literature identifies narrative-based intervention programs as effective in promoting children's SR. These interventions offer individuals the opportunity to acquire, practice, and reflect on the strategies employed by the characters to overcome their challenges. Parent participation in the Lupis program will help them transfer the content learned and associated SR strategies to their own lives, and teach them to their children. Parents' training, focused on learning SR strategies and how to teach this knowledge to their children, will be guided by the discussion of the story content following the three types of knowledge rationale: declarative, procedural, and conditional.

In addition, to improve their ability to train their children, parents will learn the SR content through the instructional sequence approach. The instructional sequence encompasses four stages: direct instruction, modeling, guided practice with feedback, and autonomous practice.

- Activities of the intervention program using the wise intervention. The main goal of a wise intervention is to help individuals (in this case, the parents) construct adaptive meanings that enable them to achieve their goals. A wise intervention is characterized by (a) short duration, (b) presentation (neither stigmatizing nor specific to clinical populations), and (c) focus (on a single belief, as opposed to many interconnected ones.

Given this, Lupis is a narrative-based, at-distance, and online intervention program based on the "Three Little Pigs" (this traditional story was chosen because it is a popular intergenerational tale known to parents and children). Lupis' structure will consist of eight weekly modules (seven modules during the first seven weeks and the last one after three months). Each module will have two moments: (1) at-distance moment with two parts: (i) parents will be presented with short reflection videos (two to five minutes each) about SR strategies (on the Edpuzzle® educational platform). The link to access will be shared in the Facebook® private groups; (ii) parents will be presented with three activities to carry out with their children; and (2) an online moment through a Zoom® session for joint reflection between parents about the content learned. Parents will be able to choose their desired level of engagement in the program, completing the minimum or all of the proposed asynchronous and synchronous steps of the intervention modules.

The investigation on the efficacy of the program will follow a cluster Randomized Controlled Trial (cRCT) design, in which elementary schools will be randomly assigned to one of the three parallel conditions: (i) Experimental Group (EG) where parents will benefit from modules about SR strategies (e.g., setting goals) through a narrative-based intervention program; (ii) Active Control Group (ACG) where parents will benefit from general educational content focusing on study methods (e.g., making a study timetable); (iii) Passive Control Group (PCG) where parents will not benefit from an intervention. Approximately 150 parents/guardians (hereinafter referred to as parents) will participate and will represent the unit of analysis for the study, and schools will be the unit of randomization.

Procedures and randomization This study was approved by the Ethics Committee for Research in Social and Humanities (CEICSH 037/2022), which can be consulted in the current study registry. The administration of the evaluation protocol for this study was also accepted by the Monitoring of Surveys in Schools (Survey No. 0461200037), coordinated by the Ministry of Education.

Elementary school boards in the north of the country will be invited to enroll in the program. Afterward, the project will be presented to teachers and parents at those schools that accept enrollment. Both parents and teachers will sign their informed consent to participate in the research (teachers will only give permission to participate in data collection). The informed consent will contain, for example: (i) a description and a timeline of the intervention program; (ii) permission to participate in data collection; (iii) as well as permission to collect data with their young children (1st and 2nd grades). However, children will also give their assent to participate in data collection after their parents have given consent for them to participate.

Therefore, each school that accepts enrollment in the program will be randomly assigned a number associated with one of the groups (i.e., EG, ACG, and PCG) on a 1:1:1 basis. Randomization will not be possible at the individual level because participants from the same class and school must be allocated to the same treatment condition to prevent contamination between groups.

Retention and incentives for the participants To promote the engagement of the parents in the intervention program and minimize their dropout, the investigators will follow good practices presented in the literature; for example, in every session, parents will be asked to check if the are any problems with their internet access, logging in to the platforms, or with their camera or audio.

In the first module, the investigators will create an introductory and welcome video, deliver guiding documents (FAQ and research team contacts), and other materials to help participants follow the Lupis program. Finally, the investigators will provide notifications and reminders in Google Calendar® and via Facebook® posts to ensure parents' awareness of module activities. Moreover, the investigators will provide feedback on the activities, promote group discussions, and include short quizzes in the Edpuzzle®.

Evaluation of the intervention program The program measures will be answered by parents (regarding their perception of PI, and their engagement in the intervention program), children (to measure SR), and teachers (regarding their perception of PI and children's use of SR strategies). All measures will be responded to at three moments of evaluation.

Statistical analysis plan Descriptive analyses will be used to characterize the sample in the treatment of sociodemographic data.

The investigators anticipate that there may be differences in the behavior of each participating parent. Thus, the analysis strategy will focus on a person-centered approach, i.e., the investigators will evaluate the impact of the intervention program by considering the clusters of participant engagement in each experimental condition (EG and ACG). Hierarchical clustering on standardized variables will be used to determine the number of clusters, followed by k-means to refine cluster fit. Intervention effects will be examined using a mixed-design ANOVA with Time (pre, post, and FUP) as a within-subject factor and Group (EG and ACG) and Cluster as between-subject factors, focusing on the Time × Group interaction and exploring the Time × Group × Cluster interaction.

A subsequent analysis will be conducted to verify if there are any natural changes over time in the PCG. To this end, a mixed-methods ANOVA with Time (pre, post, and FUP) as a within-subject factor will be conducted to examine changes over time in the PCG. All the analyses will be conducted using the IBM SPSS Statistics software.

Expected results After the person-centered analysis, distinct profiles of parents are expected to emerge within the EG and the ACG, according to their level of engagement in the intervention programs and their perception of their PI.

In the within-subjects analysis of change over time (pre - post) in each EG and ACG profile, an increase in PI and SR in children is expected. The differences found are expected to be statistically significant in each EG and ACG profile. In the FUP, it is expected that the differences found in PI and SR in children will remain stable in the EG profiles and decrease slightly in the ACG profiles (post - FUP).

In the between-subjects analysis, when comparing similar EG and ACG profiles in relation to PI and SR in children, EG profiles are expected to show a greater increase over time (pre - post). In the FUP, it is expected that the EG profiles will maintain stable the results in PI and SR in children, and in the ACG profiles, it is expected that these may decrease slightly (post - FUP). These differences are expected to be statistically significant.

As secondary outcomes, the investigators will have teachers' perceptions of PI and SR in children. In the first instance, it is expected that teachers' perceptions will increase over time (pre - post) in each EG and ACG profile. The differences found are expected to be statistically significant. In the FUP, it is expected that differences in teachers' perceptions will remain stable in the EG profiles and decrease slightly in the ACG profiles (post - FUP). Comparing teachers' perceptions of PI and SR in children in the EG and ACG profiles, it is expected that there will be a greater increase in teachers' perceptions in the EG profiles (pre - post). In the FUP, it is expected that differences in teachers' perceptions will remain stable in the EG profiles and decrease slightly in the ACG profiles (post - FUP). These differences are expected to be statistically significant.

Regarding natural changes in the PCG, no significant differences are expected over time (pre, post, and FUP) in the PI, SR in children, and teachers' perceptions of PI and SR in children.

Ethical considerations The research team declares that this project will be conducted without any commercial or financial conflicts of interest. Participants will be volunteers; no one will receive any compensation or reward for their participation, and no costs will be associated with this research. Participants with specific support needs related to health or education will be provided with alternatives delivered by entities with which the investigators have partnerships.

The evaluation protocol will not be available for consultation by anyone outside the research team. To ensure the privacy and anonymity of participants, the investigators will utilize a pseudonymization system, transforming personal data into a dataset that cannot be linked to individuals unless additional information is provided (e.g., a decoding key). These data will be stored in multiple locations, and only the principal investigator will have access to the entire dataset, which will be used solely for research purposes. Finally, all procedures for storing, processing, and protecting personal data will comply with the policies of the General Data Protection Regulation (GDPR) 2016/679; for example, all questionnaires will be destroyed five years after the end of the research. Finally, to ensure equitable access and guarantee benefits for all participants, participants in the ACG and PCG groups will be invited to enroll in the Lupis program after completing the final assessment.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children in the 1st and 2nd grades of elementary school with informed consent form;
* Parents with access to a smartphone/computer equipped with a camera and speakers;
* Parents with Internet access;
* Children with verbal consent, and parental consent;
* Teachers with informed consent.

Exclusion Criteria:

* Parents, children, and teachers who lack informed consent;
* Parents without access to the internet or an electronic device to access online content.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Parents - Sociodemographic questionnaire | Baseline (pre-intervention)
  These measures will include questions about the individuals (e.g., gender, age, level of education) and their families (e.g., number of children).
Parental Role Construction for Involvement in the Child's Education | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  This measure assesses parents' beliefs about their Involvement in the Child's Education and comprises 16 items split into two parts: (i) Part 1 (Role Activity Beliefs, ten items about parents' beliefs about what should be done in relation to their children's education, e.g., "I believe it is my responsibility to help my child with homework"). Parents will respond on a six-point Likert-like scale from 1 ("Disagree very strongly") to 6 ("Agree very strongly"); and (ii) Part 2 (Attitudes towards School, six items about parents' feelings of their school experiences when as students (e.g., "My school experience was…"). Parents will respond on a six-point Likert-like scale from 1 ("Bad") to 6 ("Good"). The Cronbach's alpha for the original was .80 and .85, respectively.
Parental Self-Efficacy for Helping the Child Succeed in School | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  This measure assesses parents' perceptions of their self-efficacy for helping the child succeed in school through seven items (e.g., "I feel successful about my efforts to help my child learn"). Parents will answer on a six-point Likert-like scale, ranging from 1 ("Disagree very strongly") to 6 ("Agree very strongly"). The Cronbach's alpha of the original study was .78.
Parents' Perceptions of Specific Invitations for Involvement from the Child | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  This measure (six items) assesses parents' perceptions of their involvement in response to their children's invitations (e.g., "My child asked me to attend a special event at school"). Parents will indicate the frequency of these invitations on a six-point Likert-like scale from 1 ("Never") to 6 ("Daily"). The Cronbach's alpha for the original study was .78.
Parents' Perceptions of Specific Invitations for Involvement from the Teacher | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  This measure (six items) assesses parents' perceptions of their involvement in response to their children's teacher invitations (e.g., "My child's teacher asked me to attend a special event at school"). Parents will indicate the frequency of these invitations on a six-point Likert-like scale from 1 ("Never") to 6 ("Daily"). The Cronbach's alpha for the original study was .81.
Parents' Perceived Life Context | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  This measure (15 items) assesses parents' perceptions of constraints (e.g., Time and Energy and Knowledge and Skills) to their involvement in the child's education. Parents will respond to the six statements about Time and Energy (e.g., "I have enough time and energy to communicate effectively with my child about the school day") and the nine statements about Knowledge and Skills (e.g., "I know enough about the subjects of my child's homework to help him or her) on a six-point Likert-like scale from 1 ("Disagree very strongly") to 6 ("Agree very strongly"). The Cronbach's alpha of the original study was .84 and .83, respectively.
Parental Involvement Mechanisms Measurement | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  This scale (51 items) assesses parents' involvement strategies and "mechanisms". Parents will respond on a six-point Likert-like scale from 1 ("Not at all true") to 6 ("Completely true") to: (i) 13 items on Encouragement (e.g., "We encourage this child to believe that he/she can learn new things"); (ii) ten items on Modeling (e.g., "We show this child that we like to learn new things"); (iii) 13 items on Reinforcement (e.g., "We show this child we like it when he or she wants to learn new things"), and (iv) 15 items on Instruction (e.g., "We teach this child to go at his or her own pace while doing schoolwork"). The Cronbach's alpha for the original study's four dimensions was .91, .88, .90, and .93, respectively.
Module assessment - engagement on platforms | During the 5-week intervention period, from baseline (pre-intervention) through immediately after the intervention (week 6)
  Parents' interactions on online platforms will be gathered as observational measures of parents' engagement in the program. The observational measures will include participants' answers to the content of the Edpuzzle® videos, comments to Facebook® posts, and the number of sessions attended on Zoom®.
Shape School | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  To assess SR strategies in children, the investigators will administer a neuropsychological test of executive functions. Shape School follows a storybook format that features cartoons with different geometric shapes (squares and circles) in various colors (red, blue, and yellow). The test consists of four experimental conditions (control, inhibition, switch, and both). The number of correctly identified stimuli and the response time are recorded for each condition, and the efficiency value is calculated by dividing the number of correct stimuli by the reaction time in each condition (Efficiency = #Correct/Total Time). The internal consistency values for Escola de Formas present an adequate result for conditions B (α = .89), C (α = .71), and D (α = .71). Except for two items, the children's answers were correct for condition A (α = 1).

SECONDARY OUTCOMES:
Teachers - sociodemographic measures | baseline (pre-intervention)
  The teachers will begin by answering brief questions about their sociodemographic data, such as their gender, age, level of education, and years of experience.
Inventory of Learning Self-regulation Processes | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  To investigate teachers' perceptions of children's use of self-regulation strategies, the investigators will adapt Inventory of Learning Self-regulation Processes (IPAA). Thus, teachers will have to answer nine adapted items based on the three phases of the SR process: (i) three items about Planning; (ii) three items about Execution; and (iii) three items about Evaluation. The teachers will evaluate the adapted items according to the frequency of observation of these parameters in the students on a five-point Likert-like scale from 1 ("Never") to 5 ("Always"). The reliability of the subscales for the original study is α = .84, α = .77, and α = .85, respectively.
School-based engagement | baseline (pre-intervention); Immediately after the intervention (6 weeks after baseline); Follow-up (3 months after the intervention; 19 weeks after baseline)
  To gather information about teachers' perceptions of PI, teachers will complete an adapted version of the School-based Engagement survey (Yamamoto et al., 2016). Thus, teachers will assess their perception of how often parents participate in their children's school activities on five items (e.g., "The parents (father and/or mother) visited in the classroom"), on a six-point Likert-like scale from 1 ("Never") to 6 ("Always"). The Cronbach's alpha of the original study was .82.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Mesquita, MSc, Principal Investigator — Psychology Research Center, School of Psychology, University of Minho, Braga, Portugal; Armanda Pereira, PhD, Study Chair — Centre for Trandisciplinary Development Studies, University of Trás-os-Montes and Alto Douro, Vila Real, Portugal.; Pedro Rosário, PhD, Study Chair — Psychology Research Center, School of Psychology, University of Minho, Braga, Portugal
Locations (1):
- University of Minho - Campus de Gualtar, Braga, Braga District, Portugal

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.

REFERENCES:
- See also: Research group website. — http://www.guia-psi.com
- See also: Facebook page of the research project. — https://www.facebook.com/profile.php?id=61562641153185
- See also: Instagram page of the research project. — https://www.instagram.com/projetolupis/